CLINICAL TRIAL: NCT04794699
Title: An Open Label, Phase 1, Treatment Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of IDE397 (MAT2A Inhibitor) In Adult Participants With Advanced Solid Tumors
Brief Title: Study of IDE397 in Participants With Solid Tumors Harboring MTAP Deletion
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: IDEAYA Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDE397-001
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2024-11

CONDITIONS: Solid Tumor
Keywords: MAT2A; 9p21; CDKN2A; MTAP; Solid Tumors; PRMT5; SAM; Synthetic Lethality; Inhibitor; MTAP deletion; CDKN2A deletion; MAT2A Inhibitor; Advanced solid tumors; Lung Cancer; Bladder Cancer; Squamous; NSCLC; Urothelial Cancer; Non small cell; Docetaxel; Paclitaxel; Sacituzumab govitecan; Trodelvy
MeSH Terms: conditions — Lung Neoplasms; Urinary Bladder Neoplasms | interventions — Docetaxel; Paclitaxel; sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1: Dose Escalation Monotherapy (Solid Tumors) (Experimental)
  Interventions: Drug: IDE397
- Part 2: Monotherapy Dose Expansion (NSCLC, EG and Urothelial) (Experimental)
  Interventions: Drug: IDE397
- Part 3: Combination Dose Escalation with docetaxel or paclitaxel (NSCLC, EG and Urothelial) (Experimental)
  Interventions: Drug: IDE397; Drug: Docetaxel; Drug: Paclitaxel
- Part 4: Combination Dose Expansion with docetaxel or paclitaxel (NSCLC, EG and Urothelial) (Experimental)
  Interventions: Drug: IDE397; Drug: Docetaxel; Drug: Paclitaxel
- Part 5: Combination Dose Escalation with sacituzumab govitecan (SG) (Urothelial) (Experimental)
  Interventions: Drug: IDE397; Drug: Sacituzumab govitecan
- Part 6: Combination Dose Expansion with sacituzumab govitecan (SG) (Urothelial) (Experimental)
  Interventions: Drug: IDE397; Drug: Sacituzumab govitecan

INTERVENTIONS:
Drug: IDE397 — IDE397 dosed orally
Drug: Docetaxel — Intravenous infusion
  Arms: Part 3: Combination Dose Escalation with docetaxel or paclitaxel (NSCLC, EG and Urothelial); Part 4: Combination Dose Expansion with docetaxel or paclitaxel (NSCLC, EG and Urothelial)
Drug: Paclitaxel — Intravenous infusion
  Arms: Part 3: Combination Dose Escalation with docetaxel or paclitaxel (NSCLC, EG and Urothelial); Part 4: Combination Dose Expansion with docetaxel or paclitaxel (NSCLC, EG and Urothelial)
Drug: Sacituzumab govitecan — Intravenous infusion
  Arms: Part 5: Combination Dose Escalation with sacituzumab govitecan (SG) (Urothelial); Part 6: Combination Dose Expansion with sacituzumab govitecan (SG) (Urothelial)

SUMMARY:
This is a Phase 1, open-label, multicenter, dose escalation and expansion study of the safety, PK, PD, and preliminary anti-tumor activity of IDE397 as a single agent and in combination with other anticancer agents including taxanes (docetaxel, paclitaxel), or sacituzumab govitecan (SG), in adult patients with selected advanced or metastatic MTAP-deleted advanced solid tumors who are unresponsive to standard of care therapy. IDE397 is a small molecule inhibitor of methionine adenosyltransferase 2 alpha (MAT2A).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18 years of age
* Advanced or metastatic solid tumor that has progressed on at least one prior line of treatment or is intolerant to additional effective standard therapy
* Have evidence of homozygous loss of MTAP or MTAP deletion
* Willing to undergo paired fresh biopsy (pre- and post-treatment) procedure. Exceptions may be made for feasibility and safety concerns
* Measurable disease
* ECOG performance status <= 1
* Adequate organ function
* Able to swallow and retain orally administered study treatment
* Recovery from acute effects of prior therapy
* Able to comply with contraceptive/barrier requirements

Exclusion Criteria:

* Known symptomatic brain metastases
* Known primary CNS malignancy
* Current active liver or biliary disease
* Impairment of gastrointestinal (GI) function
* Active uncontrolled infection
* Clinically significant cardiac abnormalities
* Previous treatment with a MAT2A inhibitor and / or PRMT inhibitor or sacituzumab govitecan
* Systemic anti-cancer therapy or major surgery within 4 weeks prior to study entry
* Radiation therapy within 2 weeks prior to study entry
* Prior irradiation to >25% of the bone marrow
* Current use or anticipated need for food or drugs that are known strong CYP3A4/5 inhibitors or inducers
* Currently receiving another investigational study drug.
* Known or suspected hypersensitivity to IDE397/excipients or components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-04-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicities (DLTs) of IDE397 | 21 days following the first dose of IDE397
  Incidence of DLTs of IDE397 will be determined
Dose-limiting Toxicities (DLTs) of IDE397 in combination with docetaxel or paclitaxel or sacituzumab govitecan | 21 - 28 days following the first dose of IDE397
  Incidence of DLTs of IDE397 in a combination setting will be determined
Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) of IDE397 | Approximately 2 years
  MTD and RP2D of IDE397 will be determined
Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) of IDE397 in combination with docetaxel or paclitaxel or sacituzumab govitecan | Approximately 2 years
  MTD and RP2D of IDE397 in a combination setting will be determined
To evaluate preliminary anti-tumor activity of IDE397 in combination expansion arms | Approximately 2 years
  Objective Response Rate (ORR) and Duration of Response (DoR)

SECONDARY OUTCOMES:
Plasma Pharmacokinetics of IDE397 and metabolite | Approximately 2 years
  Pharmacokinetics of IDE397 and metabolite following single and multiple oral administration as a single agent and in combination with docetaxel or paclitaxel or sacituzumab govitecan, will be determined
Drug interaction between IDE397 and docetaxel or paclitaxel or sacituzumab govitecan | Approximately 2 years
  Pharmacokinetics of docetaxel or paclitaxel or sacituzumab govitecan.
Pharmacodynamic effect of IDE397 as a single agent and in combination with docetaxel or paclitaxel or sacituzumab govitecan | Approximately 2 years
  Changes in the levels of MAT2A pathway and PRMT5 pathway will be determined
Preliminary anti-tumor activity in IDE397 escalation and combination escalation arms | Approximately 2 years
  Objective response rate and duration of response will be assessed by Investigator using the Response Evaluation Criteria in Solid Tumors (RECIST v1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Jasgit Sachdev, MD, Study Director — IDEAYA Biosciences
Locations (39):
- United States (20):
  - Honor Health Research Institute, Scottsdale, Arizona
  - Rockefeller Cancer Institute, Little Rock, Arkansas
  - City of Hope, Duarte, California
  - Hoag Memorial Hospital, Newport Beach, California
  - Providence Medical Group, Santa Rosa, California
  - Advent Health, Celebration, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Markey Cancer Center, Lexington, Kentucky
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Columbia University Medical Center - Herbert Irving Pavilion, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - LifeSpan - Brown University, Providence, Rhode Island
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson, Houston, Texas
  - Next Oncology, San Antonio, Texas
  - Swedish Cancer Institute, Seattle, Washington
- Australia (2):
  - The Kinghorn Cancer Centre, St Vincent's Health Network Sydney, Darlinghurst, New South Wales
  - Southern Oncology Clinical Research Unit, Bedford Park, South Australia
- France (4):
  - Institut Bergonie, Bordeaux, Bordeaux Cedex
  - Institut Claudius Regaud - IUCT-Oncopole, Toulouse, Cedex 9
  - Hôpital Timone, Marseille, Marseille
  - Centre Eugène Marquis, Rennes
- Universitaetsklinikum Hamburg-Eppendorf (UKE), Hamburg, Germany
- South Korea (5):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - CHA University - Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Sevrance Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (5):
  - Vall Hebron Institute of Oncology, Barcelona
  - Hospital Universitario 12 de Octubre (H12O), Madrid
  - START Madrid-HM - Centro Integral Oncológico Clara Campal (CIOCC), Madrid
  - NEXT Madrid, Universitary Hospital QuironSAlud, Madrid
  - Instituto Valenciano de Oncología (IVO), Valencia
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan, Tainan
  - National Taiwan University Hospital, Taipei, Taipei

IPD SHARING:
Plan to Share IPD: No